CLINICAL TRIAL: NCT06712056
Title: Effect of Mindfulness- Based Stress Reduction Program in the Elderly onSpiritual Well- Being and Meaning of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Melek Yasemin Sevimoglu, Public Health Nurse, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MYSevimoğlu
Record Dates: First submitted 2024-11-20; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Aging Well; Nursing Caries
Keywords: Mindfulness,; Nursing; Stress; Spirituality.
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: quasi-experimental study with a pretest posttest controlgroup design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm and İnterventional (Experimental): MBSR training will be given to this experimental group. To assess the cognitive status of the elderly, the "Standardized Mini-Mental State Examination" was used for those with primary or higher education levels, and the "Standardized Mini-Mental State Examination for the Uneducated" for those without primary education. Only elderly individuals scoring 23 or above on the Mini-Mental State Examination were included in the study. The elderly participants received mindfulness training (8 sessions), and personal questionnaire forms, the Spiritual Well-Being Scale, and the Meaning in Life Scale were administered before the intervention and post-intervention (at the 1st and 3rd months).The training is include awareness, staying in the moment, awareness of body, emotion, thought and environment, and breathing exercise techniques.
  Interventions: Behavioral: Mindfulness
- İnterventional (No Intervention): MBRS training will not be given to this control group

INTERVENTIONS:
Behavioral: Mindfulness — study of focusing attention
  Other Names: awereneses training; breathing awareness study.
  Arms: Arm and İnterventional

SUMMARY:
This quasi-experimental study with a pretest-posttest control group will be conducted to determine the effect of a mindfulness-based stress reduction program on spiritual well-being and the meaning of life among the elderly.

DETAILED DESCRIPTION:
Aging is a natural part of the life process, during which individuals undergo numerous biological, psychological, and social changes. In this period, people often engage in reflecting on past life experiences, seeking meaning in life, and searching for a spiritual direction. At the same time, physical limitations brought about by aging, social isolation, and losses can increase stress levels in older individuals. Stress can have adverse effects on their health, including anxiety, depression, sleep problems, and overall health deterioration.

Mindfulness-Based Stress Reduction (MBSR) helps individuals develop skills to accept the present moment, cope with stress, and regulate emotions. Spiritual well-being plays a significant role in enhancing the quality of life for older adults. The MBSR program enables older individuals to consciously focus their attention on the present moment, allowing them to live more mindfully in the "here and now" instead of dwelling on past anxieties or future worries.

This study examines the effects of the MBSR program on spiritual well-being and meaning-making in older adults, highlighting the importance of spiritual support and mindfulness practices in later life. The research aims to contribute to spiritual support programs for older individuals. A hypothesis will be tested to determine whether there is a difference between the intervention and control groups after the program's implementation.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older,

  * Living in the nursing home where the research will be conducted,
  * Being competent to continue the health education program,
  * Getting at least 23 points from SMMT
  * No hearing-visual impairment,
  * Being literate,
  * Volunteering to participate in research.

Exclusion Criteria:

* Having a communication barrier,
* Being diagnosed with dementia,
* Not having attended any session of the eight-session training program,
* Getting a score lower than 23 points from SMMT,
* Having psychosis or mental disability that may cause cognitive impairment,
* Do not have a terminal illness.
* Not having participated in any of the Pretest, Posttest-1 and Posttest-2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | pretraining
  In this study, elderly individuals, who scored at least 23 and at most 30 on the Standardized Mini Mental Test were included
Survey Form | pretraining
  The form prepared by the reseearchers consisted of 13 questions, including personal characteristics, developed based on a literature review

SECONDARY OUTCOMES:
Spiritual Well Being Scale | post-training at the 1st and 3rd months]
  The scale consists of 29 questions and three sub-dimensions with five-point Likert type items. A high score in each sub-dimensin indicats that the individual possesses the characteristic assessed by that sub-dimension. It is a three- factor scale, with a possible score range of 29 to 145.
Meaning in Life Scale | post traninig at the 1st and 3rd months
  The scale consists of 10 questions and two sub- dimensions with seven point likert type items. The correlation coefficients between the items in Turkish and original forms range from 0.65 to 0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Yasemin Sevimoğlu, Study Chair — Aydın Adnan Menderes University, Faculty of Nursing, Devision Public Health Nursing; Filiz Adana, prof, Principal Investigator — Aydın Adnan Menderes University, Faculty of Nursing, Devision Public Health Nursing
Locations (1):
- Aydın Adnan Menderes University, Faculty of Nursing, Devision Public Health Nursing, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request